CLINICAL TRIAL: NCT03575845
Title: The Effect of Yoga on Barriers to Occupational Engagement in African American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Mary University (Other)
Responsible Party: Principal Investigator, Julie H Hunley, Assistant Professor, Mount Mary University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150820
Record Dates: First submitted 2018-06-17; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Breast Neoplasm Female
Keywords: Yoga

STUDY DESIGN:
Intervention Model Description: single arm pretest-posttest design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupational therapy informed yoga (Experimental): Occupational therapists adapted postures to meet the abilities and rehabilitation needs of individual breast cancer survivors engaging in group-delivered yoga sessions
  Interventions: Behavioral: Occupational Therapy Informed Yoga

INTERVENTIONS:
Behavioral: Occupational Therapy Informed Yoga — Occupational therapy informed yoga met weekly for six, 60-minute sessions. Each session started with a seated warm-up to coordinate breath and movement and promote upper extremity mobility. Standing postures followed to target balance. Sessions closed with restorative postures in seated and supine variations.

SUMMARY:
The purpose of this study was to determine if occupational therapy informed yoga could decrease barriers to occupational engagement in African American breast cancer survivors.

.

DETAILED DESCRIPTION:
Breast cancer disproportionately affects African American women as illustrated by a 42% higher death rate and an 11% lower 5-year survival rate when compared to Caucasian women. Reasons for these disparities include biological and structural barriers to higher survival rates.

Regular physical activity and resistance training are recommended to support improved survivorship. To date, few efforts have targeted African American survivors who may experience greater survivorship challenges than Caucasians.

Yoga is a safe and effective means for breast cancer survivors to exercise and gain positive physical and psychosocial outcomes. Only two studies, 10 years apart, have provided evidence about the efficacy of yoga for African American breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* Breast Cancer survivor
* No medical restrictions on activity

Exclusion Criteria:

* Race other than African American
* No history of breast cancer
* Medical restrictions on activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2015-07-16 (Actual); Study Completion 2015-10-24 (Actual)

PRIMARY OUTCOMES:
Change in dynamic balance | Week 1 & week 6
  Dynamic balance measured with Functional Reach Assessment

SECONDARY OUTCOMES:
Change in Pain | Week 1 & week 6
  Universal Pain Assessment Tool
Change in Mental Health | Week 1 & week 6
  Mental health subscale of Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Julie H Hunley, PhD, Principal Investigator — Mount Mary University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moadel AB, Shah C, Wylie-Rosett J, Harris MS, Patel SR, Hall CB, Sparano JA. Randomized controlled trial of yoga among a multiethnic sample of breast cancer patients: effects on quality of life. J Clin Oncol. 2007 Oct 1;25(28):4387-95. doi: 10.1200/JCO.2006.06.6027. Epub 2007 Sep 4. PMID 17785709
- [Background] Taylor TR, Barrow J, Makambi K, Sheppard V, Wallington SF, Martin C, Greene D, Yeruva SLH, Horton S. A Restorative Yoga Intervention for African-American Breast Cancer Survivors: a Pilot Study. J Racial Ethn Health Disparities. 2018 Feb;5(1):62-72. doi: 10.1007/s40615-017-0342-4. Epub 2017 Apr 14. PMID 28411330
- [Background] Daly B, Olopade OI. A perfect storm: How tumor biology, genomics, and health care delivery patterns collide to create a racial survival disparity in breast cancer and proposed interventions for change. CA Cancer J Clin. 2015 May-Jun;65(3):221-38. doi: 10.3322/caac.21271. Epub 2015 Apr 9. PMID 25960198
- [Background] Coughlin SS, Yoo W, Whitehead MS, Smith SA. Advancing breast cancer survivorship among African-American women. Breast Cancer Res Treat. 2015 Sep;153(2):253-61. doi: 10.1007/s10549-015-3548-3. Epub 2015 Aug 25. PMID 26303657
- [Background] Mollica M, Newman SD. Breast cancer in African Americans: from patient to survivor. J Transcult Nurs. 2014 Oct;25(4):334-40. doi: 10.1177/1043659614524248. Epub 2014 Mar 4. PMID 24595162
- [Background] Bower JE, Garet D, Sternlieb B, Ganz PA, Irwin MR, Olmstead R, Greendale G. Yoga for persistent fatigue in breast cancer survivors: a randomized controlled trial. Cancer. 2012 Aug 1;118(15):3766-75. doi: 10.1002/cncr.26702. Epub 2011 Dec 16. PMID 22180393
- [Background] Harder H, Parlour L, Jenkins V. Randomised controlled trials of yoga interventions for women with breast cancer: a systematic literature review. Support Care Cancer. 2012 Dec;20(12):3055-64. doi: 10.1007/s00520-012-1611-8. Epub 2012 Oct 6. PMID 23052917
- [Background] Littman AJ, Bertram LC, Ceballos R, Ulrich CM, Ramaprasad J, McGregor B, McTiernan A. Randomized controlled pilot trial of yoga in overweight and obese breast cancer survivors: effects on quality of life and anthropometric measures. Support Care Cancer. 2012 Feb;20(2):267-77. doi: 10.1007/s00520-010-1066-8. Epub 2011 Jan 5. PMID 21207071
- [Background] Levine AS, Balk JL. Yoga and quality-of-life improvement in patients with breast cancer: a literature review. Int J Yoga Therap. 2012;(22):95-9. PMID 23070679